CLINICAL TRIAL: NCT04135989
Title: Randomized 2x2 Factorial Trial Comparing the Cre8 Amphilimus-sirolimus Eluting Stent vs. the Synergy Everolimus-eluting Stent and a Personalized vs. Standard Duration of Dual Antiplatelet Therapy in All-comers Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Personalized Vs. Standard Duration of Dual Antiplatelet Therapy and New-generation Polymer-Free vs- Biodegradable-Polymer DES
Acronym: PARTHENOPE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: AdvicePharma Group (Unknown)
Responsible Party: Principal Investigator, Giovanni Esposito, Professor of Cardiology, Federico II University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 197/19
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Chronic Coronary Syndrome; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: 2-by-2 randomization
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cre8 AES and personalized DAPT duration (Other): Percutaneous coronary intervention with implantation of a Cre8 amphilimus- eluting stent for coronary artery disease.
  Personalized duration of dual antiplatelet therapy for 3-, 6-, or 24-month after percutaneous coronary intervention based on the DAPT score.
  Interventions: Device: Percutaneous coronary intervention with implantation of amphilimus-eluting stents for coronary artery disease.; Drug: Personalized DAPT duration
- Cre8 AES and standard DAPT duration (Other): Percutaneous coronary intervention with implantation of a Cre8 amphilimus- eluting stent for coronary artery disease.
  Standard duration of dual antiplatelet therapy for 12-month after percutaneous coronary intervention.
  Interventions: Device: Percutaneous coronary intervention with implantation of amphilimus-eluting stents for coronary artery disease.; Drug: Standard DAPT duration
- Synergy EES and personalized DAPT duration (Other): Percutaneous coronary intervention with implantation of a Synergy everolimus-eluting stent for coronary artery disease.
  Personalized duration of dual antiplatelet therapy for 3-, 6-, or 24-month after percutaneous coronary intervention based on the DAPT score.
  Interventions: Device: Percutaneous coronary intervention with implantation of everolimus-eluting stents for coronary artery disease.; Drug: Personalized DAPT duration
- Synergy EES and standard DAPT duration (Other): Percutaneous coronary intervention with implantation of a Synergy everolimus-eluting stent for coronary artery disease.
  Standard duration of dual antiplatelet therapy for 12-month after percutaneous coronary intervention.
  Interventions: Device: Percutaneous coronary intervention with implantation of everolimus-eluting stents for coronary artery disease.; Drug: Standard DAPT duration

INTERVENTIONS:
Device: Percutaneous coronary intervention with implantation of amphilimus-eluting stents for coronary artery disease. — Implantation of polymer-free, amphilimus-eluting, drug-eluting stents
  Other Names: Cre8 AES
  Arms: Cre8 AES and personalized DAPT duration; Cre8 AES and standard DAPT duration
Device: Percutaneous coronary intervention with implantation of everolimus-eluting stents for coronary artery disease. — Implantation of biodegradable-polymer, everolimus-eluting, drug-eluting stents
  Other Names: Synergy EES
  Arms: Synergy EES and personalized DAPT duration; Synergy EES and standard DAPT duration
Drug: Personalized DAPT duration — Duration of dual antiplatelet therapy according to DAPT score for 3- or 6- months in patients with low DAPT score (stable CAD or ACS, respectively) or for 24-months in patients with high DAPT score
  Arms: Cre8 AES and personalized DAPT duration; Synergy EES and personalized DAPT duration
Drug: Standard DAPT duration — Duration of dual antiplatelet therapy for 12 months.
  Arms: Cre8 AES and standard DAPT duration; Synergy EES and standard DAPT duration

SUMMARY:
New-generation metallic drug-eluting stents represent the standard of care among patients undergoing percutaneous coronary intervention (PCI). Currently, few data are available as regards to the safety and efficacy of the Cre8 amphilimus-eluting stent (Cre8 AES, Alvimedica, Instanbul, Turkey) in comparison with the biodegradable polymer everolimus-eluting stent (Synergy EES, Boston Scientific, Marlborough, MA, USA). Results from randomized trials and meta-analyses consistently indicate that prolonged dual antiplatelet therapy (DAPT) after PCI reduces ischemic events, but invariably conveys an excess of clinically relevant bleeding, which is proportional to the duration of treatment. It has been estimated, indeed, that for every non-fatal ischemic event avoided with prolonged DAPT, two or more clinically relevant bleeding events have to be expected. Given the trade-off between benefits and risks and the lack of mortality benefit in favor of prolonged DAPT, expert consensus suggests that DAPT duration should be individualized based on ischemic versus bleeding risks. At this regard, the DAPT score has been recently proposed as standardized tool to identify patients who derive benefit or lack from a prolonged course of DAPT. However, a prospective assessment of the DAPT score is lacking and whether a personalized duration of DAPT based on the DAPT score improves the net clinical benefit remains unknown.

The objective of the study is to compared the safety and the efficacy of the Cre8 AES with the Synergy EES and a personalized DAPT duration based on the DAPT score with a standard DAPT duration among patients undergoing PCI.

DETAILED DESCRIPTION:
The objective of the trial is:

i) to evaluate the efficacy and safety of the Cre8 AES vs. the Synergy EES in a broadly unselected patient population with coronary artery disease undergoing PCI; ii) to compare the safety and efficacy of a personalized DAPT duration (3-, 6-, or 24-month) guided by the application of the DAPT score with a standard DAPT duration (12-month) after PCI.

In particular, the objectives of the trial are to test the following hypothesis:

* The Cre8 AES is non-inferior to the Synergy EES with regards to a device-oriented composite endpoint (DOCE) at 1-year follow-up.
* A personalized DAPT duration based on the DAPT score is superior to a standard DAPT duration with regards to a net adverse clinical endpoint (NACE) at 2-year follow-up.

This is a prospective, randomized, multicenter, investigator-initiated, assessor-blind trial to be conducted at interventional cardiology centers in Italy. Patients undergoing PCI will be randomized in a 2-by-2 randomization fashion to undergo PCI with the Cre8 AES or Synergy EES and to receive a personalized or standard DAPT duration. All patients will be followed at 3-, 6-, 12- and 24-month after PCI for clinical endpoints.

Use of experimental and control DES:

Both the study stent (Cre8 AES) and the control stent (Synergy EES) will be used according to their indications for use. The randomly assigned stent is not expected to have an influence on the conduct of the procedure that will take place according to the routine practice. Eligible patients will undergo PCI as per local protocol, according to current guidelines of the European Society of Cardiology on myocardial revascularization. The technique of PCI (vascular access route, choice of the vascular sheath diameter, choice of the diagnostic and guiding catheters sizes and shapes, choice of the coronary guidewire) will be left to the discretion of the operator as per standard individual and local practice. The operator will choose the appropriate length and diameter of the stents to be implanted by visual estimate or quantitative coronary angiography as per local practice. The Cre8 AES and the Synergy EES systems are commercially available and all sizes may be used for the study.

DAPT duration according to randomization:

DAPT duration in patients randomized to personalized DAPT regimen: In patients that are randomized to a personalized DAPT and have a low DAPT score (<2), DAPT duration is recommended for 3 months in case of stable coronary artery disease at the time of the index procedure or for 6 months in case of acute coronary syndrome at the time of the index procedure. A low dose of aspirin (75 to 162 mg daily) will be administered throughout the course of the study. In patients that are randomized to a personalized DAPT and have a high DAPT score (≥2), DAPT duration is recommended for 24 months. Changes in the dose or in the type of P2Y12 receptor inhibitor (clopidogrel, prasugrel, or ticagrelor) are allowed during the course of the study. A low dose of aspirin (75 to 162 mg daily) will be administered throughout the course of the study. At 12-month, patients on treatment with prasugrel or ticagrelor should continue the same P2Y12 receptor inhibitor. In this specific scenario, it is preferable to continue with the same P2Y12 receptor inhibitor (prasugrel 10 mg daily or ticagrelor 90 mg daily) or to switch to a low-dose regimen of ticagrelor (60 mg twice daily) if clinically indicated or to switch to clopidogrel (75 mg daily).

DAPT regimen in patients in patients randomized to a standard DAPT duration: In patients that are randomized to a standard DAPT duration, oral P2Y12 inhibitors (clopidogrel, prasugrel, or ticagrelor) should be administered for 12-month. A low dose of aspirin (75 to 162 mg daily) will be administered throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Clinical evidence of coronary artery disease requiring PCI with DES implantation;
3. Any coronary lesion sized 2.25-4.5 mm by visual estimation.

Exclusion Criteria:

1. Inability to provide informed consent;
2. Active bleeding requiring medical attention (BARC ≥2);
3. Need for chronic oral anticoagulant therapy;
4. Planned surgery within 3 months;
5. Known hypersensitivity or allergy to aspirin or any P2Y12 receptor inhibitor (clopidogrel, prasugrel, ticagrelor), heparin, contrast agent, or any DES-components;
6. Previous treatment with bioresorbable vascular scaffolds;
7. Participation in another study that has not reached the primary endpoint;
8. A life expectancy of less than 24 months;
9. Female of childbearing potential;
10. Under judicial protection, tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2106 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2024-10-24 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Device-oriented composite endpoint (DOCE) for the comparison between the Cre8 AES and the Synergy EES. | 12 months
  The composite of cardiovascular death, myocardial infarction not clearly attributable to a non-target vessel, or clinically-driven target-lesion revascularization.
Number of Participants with Net adverse clinical endpoint (NACE) for the comparison between a personalized and standard DAPT duration. | 24 months
  The composite of all-cause death, any myocardial infarction, stroke, urgent target-vessel revascularization, or BARC type 2 to 5 bleeding at 24-month follow-up.

SECONDARY OUTCOMES:
Number of Participants with All-cause death | 12- and 24-month
Number of Participants with Death from cardiovascular causes | 12- and 24-month
Number of Participants with Myocardial infarction | 12- and 24-month
Number of Participants with Stroke | 12- and 24-month
Number of Participants with Clinically-driven target-lesion revascularization | 12- and 24-month
Number of Participants with Definite or probable stent thrombosis | 12- and 24-month
Number of Participants with Definite stent thrombosis | 12- and 24-month
Number of Participants with Any revascularization | 12- and 24-month
Number of Participants with Clinically-driven target-vessel revascularization | 12- and 24-month
Number of Participants with Urgent target-vessel revascularization | 12- and 24-month
Number of Participants with Urgent non-target-vessel revascularization | 12- and 24-month
Number of Participants with Any target-lesion revascularization | 12- and 24-month
Number of Participants with Any target-vessel revascularization | 12- and 24-month
Number of Participants with Bleeding events | 12- and 24-month
  Bleeding events according to the BARC, TIMI and GUSTO classification

CONTACTS AND LOCATIONS:
Locations (13):
- Italy (13):
  - Casa di Cura Villa Dei Fiori, Acerra, Naples
  - Ospedale S.Maria delle Grazie, Pozzuoli, Naples
  - Ospedale "Maria SS. Addolorata", Eboli, SA
  - A.O.R.N. S.Giuseppe Moscati-Città Ospedaliera, Avellino
  - Ospedale San Giuseppe Moscati, Aversa
  - A.O.R.N. Sant'Anna e San Sebastiano, Caserta
  - Ospedale San Giuliano, Giugliano in Campania
  - Federico II University of Naples, Naples
  - A.O.R.N. A. Cardarelli, Napoli
  - Ospedale San Giovanni Bosco - ASL Napoli 1, Napoli
  - Ospedale del Mare, Napoli
  - Ospedale Santa Maria della Pietà, Nola
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Piccolo R, Windecker S. Dual Antiplatelet Therapy in Percutaneous Coronary Intervention: A Tale of 2 Decades With New Perspectives in the Era of New-Generation Drug-Eluting Stents. Circ Cardiovasc Interv. 2016 Feb;9(2):e003587. doi: 10.1161/CIRCINTERVENTIONS.116.003587. No abstract available. PMID 26858081
- [Background] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- [Background] Spencer FA, Prasad M, Vandvik PO, Chetan D, Zhou Q, Guyatt G. Longer- Versus Shorter-Duration Dual-Antiplatelet Therapy After Drug-Eluting Stent Placement: A Systematic Review and Meta-analysis. Ann Intern Med. 2015 Jul 21;163(2):118-26. doi: 10.7326/M15-0083. PMID 26005909
- [Background] Bittl JA, Baber U, Bradley SM, Wijeysundera DN. Duration of Dual Antiplatelet Therapy: A Systematic Review for the 2016 ACC/AHA Guideline Focused Update on Duration of Dual Antiplatelet Therapy in Patients With Coronary Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2016 Sep 6;68(10):1116-39. doi: 10.1016/j.jacc.2016.03.512. Epub 2016 Mar 29. PMID 27036919
- [Background] Levine GN, Bates ER, Bittl JA, Brindis RG, Fihn SD, Fleisher LA, Granger CB, Lange RA, Mack MJ, Mauri L, Mehran R, Mukherjee D, Newby LK, O'Gara PT, Sabatine MS, Smith PK, Smith SC Jr. 2016 ACC/AHA Guideline Focused Update on Duration of Dual Antiplatelet Therapy in Patients With Coronary Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2016 Sep 6;68(10):1082-115. doi: 10.1016/j.jacc.2016.03.513. Epub 2016 Mar 29. No abstract available. PMID 27036918
- [Background] Raber L, Piccolo R. CardioPulse: Different bleeding scores and which one should we use? Eur Heart J. 2016 Jan 21;37(4):327-31. No abstract available. PMID 27462674
- [Background] Yeh RW, Secemsky EA, Kereiakes DJ, Normand SL, Gershlick AH, Cohen DJ, Spertus JA, Steg PG, Cutlip DE, Rinaldi MJ, Camenzind E, Wijns W, Apruzzese PK, Song Y, Massaro JM, Mauri L; DAPT Study Investigators. Development and Validation of a Prediction Rule for Benefit and Harm of Dual Antiplatelet Therapy Beyond 1 Year After Percutaneous Coronary Intervention. JAMA. 2016 Apr 26;315(16):1735-49. doi: 10.1001/jama.2016.3775. PMID 27022822
- [Background] Piccolo R, Gargiulo G, Franzone A, Santucci A, Ariotti S, Baldo A, Tumscitz C, Moschovitis A, Windecker S, Valgimigli M. Use of the Dual-Antiplatelet Therapy Score to Guide Treatment Duration After Percutaneous Coronary Intervention. Ann Intern Med. 2017 Jul 4;167(1):17-25. doi: 10.7326/M16-2389. Epub 2017 Jun 13. PMID 28605779
- [Background] Rozemeijer R, Stein M, Voskuil M, van den Bor R, Frambach P, Pereira B, Koudstaal S, Leenders GE, Timmers L, Rittersma SZ, Kraaijeveld AO, Agostoni P, Roes KC, Doevendans PA, Stella PR; ReCre8 Study Investigators. Randomized All-Comers Evaluation of a Permanent Polymer Zotarolimus-Eluting Stent Versus a Polymer-Free Amphilimus-Eluting Stent. Circulation. 2019 Jan 2;139(1):67-77. doi: 10.1161/CIRCULATIONAHA.118.037707. PMID 30586704
- [Background] Navarese EP, Andreotti F, Schulze V, Kolodziejczak M, Buffon A, Brouwer M, Costa F, Kowalewski M, Parati G, Lip GY, Kelm M, Valgimigli M. Optimal duration of dual antiplatelet therapy after percutaneous coronary intervention with drug eluting stents: meta-analysis of randomised controlled trials. BMJ. 2015 Apr 16;350:h1618. doi: 10.1136/bmj.h1618. PMID 25883067
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620
- [Derived] Piccolo R, Calabro P, Carrara G, Simonetti F, Varricchio A, Attisano T, Napolitano G, De Simone C, Carpinella G, Stabile E, Cirillo P, Di Serafino L, Caiazzo G, Tesorio T, Boccalatte M, Tuccillo B, Avvedimento M, Leone A, Galasso G, Cesaro A, Perrotta R, Niglio T, Castiello DS, Immobile Molaro M, Bardi L, Spinelli A, Cristiano S, Bellino M, Leonardi S, Biscaglia S, Costa F, Cassese S, McFadden E, Heg D, Stefanini GG, Franzone A, Capodanno D, Esposito G; PARTHENOPE Study Group. Personalized or Standard Duration of Dual Antiplatelet Therapy After Percutaneous Coronary Intervention: The PARTHENOPE Randomized Trial. J Am Coll Cardiol. 2025 Dec 9;86(23):2352-2367. doi: 10.1016/j.jacc.2025.08.040. Epub 2025 Aug 30. PMID 40892607
- [Derived] Piccolo R, Calabro P, Carrara G, Varricchio A, Baldi C, Napolitano G, De Simone C, Mauro C, Stabile E, Caiazzo G, Tesorio T, Boccalatte M, Tuccillo B, Cirillo P, Di Serafino L, Simonetti F, Leone A, Angellotti D, Bottiglieri G, Russolillo E, Galasso G, Perrotta R, Cesaro A, Niglio T, Capasso M, Spinelli A, Cristiano S, Faretra A, Bruzzese D, Chieffo A, Tarantini G, Leonardi S, Biscaglia S, Costa F, Cassese S, McFadden E, Heg D, Franzone A, Stefanini GG, Capodanno D, Esposito G, Parthenope Investigators FT. Polymer-free versus biodegradable-polymer drug-eluting stent in patients undergoing percutaneous coronary intervention: an assessor-blind, non-inferiority, randomised controlled trial. EuroIntervention. 2025 Jan 6;21(1):58-72. doi: 10.4244/EIJ-D-24-00657. PMID 39773824
- [Derived] Piccolo R, Calabro P, Varricchio A, Baldi C, Napolitano G, De Simone C, Mauro C, Stabile E, Caiazzo G, Tesorio T, Boccalatte M, Tuccillo B, Bottiglieri G, Russolillo E, Di Lorenzo E, Carrara G, Cassese S, Leonardi S, Biscaglia S, Costa F, McFadden E, Heg D, Franzone A, Stefanini GG, Capodanno D, Esposito G. Rationale and design of the PARTHENOPE trial: A two-by-two factorial comparison of polymer-free vs biodegradable-polymer drug-eluting stents and personalized vs standard duration of dual antiplatelet therapy in all-comers undergoing PCI. Am Heart J. 2023 Nov;265:153-160. doi: 10.1016/j.ahj.2023.08.001. Epub 2023 Aug 10. PMID 37572785